CLINICAL TRIAL: NCT00449202
Title: A Phase 2a Randomized, Double-Blind, Placebo Controlled, Parallel Group, Safety and Efficacy Study of Two 14 Day Cycles of Oral Doses of Oleoyl-Estrone (MP-101) in Obese Adult Subjects
Brief Title: Phase 2a Obesity Study of Oral Doses of Oleoyl-Estrone (MP-101)
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Manhattan Pharmaceuticals (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MAN-OE-OS-03
Expanded Access: Available
Record Dates: First submitted 2007-03-16; First posted 2007-03-20 (Estimated); Last update posted 2007-03-20 (Estimated); Status verified 2007-03

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity | interventions — oleoyl-estrone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: oleoyl-estrone (MP 101)

SUMMARY:
The purpose of this study is to evaluate the safety, preliminary efficacy, and pharmacokinetics of two 14-day cycles of escalating oral doses of MP 101 in 100 obese adult subjects.

ELIGIBILITY:
Inclusion Criteria:

* Be a male or female between the ages of 18 and 65 years, inclusive
* Female subjects must be either surgically sterile or at least 2 years postmenopausal
* Have a BMI of 27 - 38.9, inclusive
* Have a stable weight for the past 30 days per subject report
* Be otherwise healthy and have an acceptable medical history
* Have negative urinalysis test results for drugs of abuse and alcohol
* Have the ability to understand the requirements of the study, have provided written informed consent and agree to abide by the study restrictions
* Exhibit stable behavior patterns with regard to smoking and exercise
* Subject who has at least one factor of the metabolic syndrome

Exclusion Criteria:

* Be pregnant or nursing
* Have taken exclusionary medication in the past 30 days
* Have any clinically significant abnormal laboratory test as determined by the investigator
* Have a clinically significant illness during the 30 days before enrollment
* Have a history of testing positive for Hepatitis B virus, Hepatitis C virus, or HIV
* Have a confirmed diagnosis or history of cancer, with the exception of nonmelanoma skin cancer
* Have a previous diagnosis of diabetes
* Be otherwise unsuitable for the study, in the opinion of the investigator
* Have an allergy to safflower seeds or its byproducts (e.g., safflower oil)
* Have any postmenopausal bleeding within the last 6 months
* Have been involved in a formal or informal (self-imposed) diet regimen within the last 30 days
* Currently working night shifts
* Have a history of known multiple miscarriages

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100
Dates: Start 2006-06

PRIMARY OUTCOMES:
To evaluate the safety and tolerability

SECONDARY OUTCOMES:
To evaluate the preliminary efficacy

CONTACTS AND LOCATIONS:
Locations (3):
- United States (2):
  - Pennington Biomedical Research, Baton Rouge, Louisiana
  - Jean Brown Research, Salt Lake City, Utah
- Swiss Pharma Contract, Basel, Switzerland